CLINICAL TRIAL: NCT07374354
Title: Assessment of Preemptive/Preoperative Analgesia Effect on Pain Perception and Anxiety Management in Children With Molar Incisor Hypo-Mineralization During Restorative Treatment of First Permanent Molar: A Triple-Blinded Randomized Clinical Trial.
Brief Title: Preemptive Analgesia for Pain and Anxiety Control in Children With MIH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Esraa Diaaeldin Nady Elhenie, general practitioner, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Esraa MSA University
Record Dates: First submitted 2025-11-23; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pain and Anxiety in Children With MIH
Keywords: Molar Incisor Hypomineralization (MIH); Preemptive Analgesia; Ibuprofen; Dental Pain; Dental Anxiety; FLACC Scale; Wong-Baker FACES; Post-Eruptive Enamel Breakdown; Children 6-12 Years; Analgesic Efficacy
MeSH Terms: conditions — Pain; Molar Hypomineralization; Toothache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ibuprofen 100mg/ml oral suspension syrup (Experimental): The analgesic will be labeled A; (ibuprofen 100 mg/ml oral suspension). Administration of analgesic will be 30 mins prior to procedure.
  The Operator who will perform the restorative treatment, the participant, and their guardian will not know which suspension will be administered (analgesic or placebo) or who analyzed the data. Only the professional who will administer the drug or placebo to the child and an external dental professional will know which will be used for each child, in case of any complications during the procedure.
  Local anesthesia administration using 1.8-mL of articaine 4% with epinephrine 1:100000.
  Rubber dam will be applied, then defect removal and cavity preparation and restorative treatment will be established.
  Interventions: Drug: ibuprofen 100mg/ml oral suspension syrup
- placebo (Placebo Comparator): The placebo will be labeled B and will be sharing the same characteristics and flavor as the analgesic. Administration of placebo will be 30 mins prior to procedure.
  The Operator who will perform the restorative treatment, the participant, and their guardian will not know which suspension will be administered (analgesic or placebo) or who analyzed the data. Only the professional who will administer the drug or placebo to the child and an external dental professional will know which will be used for each child, in case of any complications during the procedure.
  Local anesthesia administration using 1.8-mL of articaine 4% with epinephrine 1:100000.
  Rubber dam will be applied, then defect removal and cavity preparation and restorative treatment will be established.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ibuprofen 100mg/ml oral suspension syrup — ibuprofen 100 mg/ml oral suspension administration 30 mins prior to procedure to assess the effect of preemptive analgesia on pain perception and anxiety management during restorative treatment of first permanent molars in children with molar incisor hypo-mineralization affected molars.
  Arms: ibuprofen 100mg/ml oral suspension syrup
Drug: Placebo — the placebo will be labeled B and will be sharing the same characteristics and flavor as the analgesic. Administration placebo will be 30 mins prior to procedure to assess the effect of preemptive analgesia on pain perception and anxiety management during restorative treatment of first permanent molars in children with molar incisor hypo-mineralization affected molars.
  Arms: placebo

SUMMARY:
This randomized, triple-blinded clinical trial aims to evaluate the effect of preemptive analgesia using ibuprofen on pain perception and anxiety during restorative treatment of first permanent molars in children diagnosed with molar-incisor hypomineralization (MIH). MIH-affected teeth often present with hypersensitivity, difficulty in achieving adequate anesthesia, and increased dental anxiety, which complicates dental treatment. Participants aged 6-12 years with MIH will receive either ibuprofen syrup or placebo 30 minutes before treatment. Pain will be assessed using the FLACC Behavioral Pain Scale and Wong-Baker FACES scale, and anxiety will be evaluated through heart rate and oxygen saturation. The results will determine whether preoperative ibuprofen reduces intraoperative pain and improves anxiety control in this population.

DETAILED DESCRIPTION:
Molar-incisor hypomineralization (MIH) is a developmental enamel defect associated with post-eruptive breakdown, hypersensitivity, difficulty achieving effective anesthesia, increased dental anxiety, and a higher risk of restorative complications. Children with MIH require more frequent and complex dental care and often experience discomfort during treatment, negatively impacting their cooperation and oral-health-related quality of life.

Preemptive analgesia-the administration of analgesics before starting dental procedures-has shown promise in reducing nociceptive transmission and improving anesthetic efficacy. Previous studies have evaluated the effect of ibuprofen on pain during dental procedures in MIH-affected children, but evidence remains limited, and anxiety-related outcomes have not been comprehensively assessed.

This triple-blinded randomized controlled trial will include children aged 6-12 presenting with MIH and post-eruptive enamel breakdown but without carious lesions or prior restorations. Participants will be randomly assigned (1:1) to receive either ibuprofen 100 mg syrup or a matching placebo 30 minutes before treatment. All procedures will be performed under standardized conditions, including local anesthesia with articaine 4%, rubber dam isolation, and restorative treatment by trained pediatric dentists.

Pain perception will be recorded using both objective and subjective metrics. Objective pain will be evaluated using the FLACC Behavioral Pain Scale during anesthesia and treatment. Subjective pain will be assessed using the Wong-Baker FACES scale at predefined time points before, during, and after treatment. Dental anxiety will be monitored using physiological indicators: heart rate and oxygen saturation measured with a pulse oximeter at baseline, during, and after the dental procedure.

The primary objective is to determine whether preemptive ibuprofen reduces behavioral pain responses during treatment. Secondary objectives include assessing self-reported pain and physiologic anxiety measures. The findings aim to guide pediatric clinicians in improving pain control, reducing treatment-related anxiety, and enhancing the overall management of children with MIH.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with molar incisor hypo-mineralization.
2. Patient's age ranges from 6 to 12 years old.
3. The affected tooth has demarcated opacity with post eruptive enamel breakdown.
4. No cavitated lesion is related to the defect of previous restorative or preventive treatment.

Exclusion Criteria:

1. Children who are physically or mentally disabled or having any medical condition that will affect or complicate assessment of the intervention.
2. Loss of tooth structure due to caries.
3. intolerance to ibuprofen.
4. developmental defects, including amelogenesis imperfecta and dentinogenesis imperfecta.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception (objective) | during injection and during procedure
  Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Pain Scale. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
pain perception (subjective) | Initial before procedure (baseline) After drug/placebo administration (30 min), Before anesthesia, After anesthesia, During the procedure (real-time) 24 hours after the end of the procedure (post-operative)
  Wong Baker FACES Pain Rating Scale. It consists of several faces ranging from happy (0) to crying (10).
dental anxiety | initial before treatment (baseline), during anesthesia, during treatment (real-time) and immediately after treatment (post-operative)
  pulse oximeter (heart rate monitor) unit: Beat/ minute
dental anxiety | initial before treatment (baseline), during anesthesia, during treatment (real-time) and immediately after treatment (post-operative)
  pulse oximeter oxygen saturation unit: percentage

CONTACTS AND LOCATIONS:
Locations (1):
- October university of modern science and arts, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes